CLINICAL TRIAL: NCT06971107
Title: TKRCD-MSI Study: Current Microsatellite Stability Findings in Colon Cancer - Nationwide Experience From Turkey
Brief Title: Current Microsatellite Stability Results in Colon Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Turkish Society of Colon and Rectal Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: TKRCD-MSI
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Colon Adenocarcinoma; MSI Positive Colorectal Cancer; MSI Negative Colorectal Cancer
Keywords: Colorectal Neoplasms; Microstaellite Instability; DNA Mismatch Repair; Immunohistochemistry; Prognosis; Survival Analysis; Epidemiologic Methods
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MLH1/PMS2 loss group: Participants whose tumors show loss of MLH1 and PMS2 protein expression, typically associated with dMMR or MLH1 promoter hypermethylation. These tumors will be analyzed for clinical features and oncologic outcomes (DFS and OS) over 3 years.
- MSH2/MSH6 Loss Group: Participants whose tumors show loss of MSH2 and MSH6 protein expression. This pattern is commonly associated with Lynch syndrome, a hereditary form of mismatch repair deficiency. Prognostic and treatment outcome data will be analyzed.
- Sporadic Group (pMMR): Participants with no loss of MMR protein expression (proficient MMR; pMMR). These cases represent sporadic tumors without mismatch repair deficiency and will serve as a comparison group for evaluating oncologic outcomes.

SUMMARY:
The goal of this prospective observational study is to learn more about how a specific type of DNA repair issue-called mismatch repair deficiency (dMMR)-affects colon cancer in people living in Turkey. The study will look at how often dMMR occurs, how it is reported, and how it relates to treatment outcomes.

The main questions it aims to answer are:

* How common is dMMR in colon cancer, and does it vary by where the tumor is in the colon?
* How often is MSI (microsatellite instability) status reported in colon cancer biopsy reports before surgery?
* How do different types of dMMR (such as MLH1/PMS2 loss, MSH2/MSH6 loss, or sporadic cases) affect survival over three years?

Participants will:

* Be people who had surgery for colon cancer between June 1, 2025 and May 31, 2026 at hospitals in Turkey that treat more than 30 colon cancer cases each year.
* Have their medical and pathology data reviewed, including information about tumor location, biopsy results, surgery, and treatment.

This study will not involve any new treatments. Instead, it will use existing medical records to better understand how to improve care and identify people who may benefit from immunotherapy. Results from this study will be shared at scientific meetings and published in medical journals.

DETAILED DESCRIPTION:
This is a prospective, multicenter observational study designed to evaluate the distribution and clinical relevance of microsatellite instability (MSI) and mismatch repair (MMR) subtypes in patients undergoing curative colon cancer surgery across Turkey. The study will run between June 1, 2025, and May 31, 2026, and is being conducted to address gaps in national data on MSI frequency and subtype patterns, which have critical prognostic and therapeutic implications.

Mismatch repair deficiency (dMMR) leads to genetic instability and is commonly associated with high levels of microsatellite instability (MSI-H). This condition results from the loss of expression in key MMR proteins-MLH1, PMS2, MSH2, and MSH6-and is linked to distinct tumor behaviors, including:

* Improved overall survival compared to MMR-proficient tumors
* Reduced risk of nodal and distant metastases
* Increased resistance to 5-fluorouracil (5-FU) and potential sensitivity to oxaliplatin
* Favorable response to immune checkpoint inhibitors, including neoadjuvant immunotherapy in selected patients with MSI-H/dMMR tumors

The primary objective of this study is to determine the prevalence and anatomical distribution of dMMR in colon cancer.

The secondary objective is to assess how frequently MSI status is reported in preoperative endoscopic biopsies.

The tertiary objective is to compare 3-year disease-free survival (DFS) and overall survival (OS) across three subtypes:

* MLH1/PMS2 loss
* MSH2/MSH6 loss
* Sporadic cases

Study Procedures:

Participating Centers:

Hospitals with an annual volume of >30 curative colon cancer surgeries will be invited to participate. Each center will assign a local principal investigator and sign a collaboration agreement.

Data Collection:

Demographic, clinical, surgical, histopathological, and molecular data will be collected. Specific variables include:

* Age, sex
* Clinical TNM stage
* Tumor size and location
* MSI status in both biopsy and resection specimens
* Neoadjuvant treatment details
* Histologic subtype and grade
* Number of retrieved and metastatic lymph nodes
* Presence of lymphatic, perineural, and venous invasion
* Tumor budding
* Immunohistochemical expression of MMR proteins (MLH1, PMS2, MSH2, MSH6)

Eligibility:

* Inclusion Criteria:
* Signed informed consent
* Undergoing curative colon cancer surgery between study dates
* Routine MSI reporting available on biopsy and/or surgical specimens
* Exclusion Criteria:
* Non-adenocarcinoma malignancies of the colon
* Rectal cancers

Sample Size Assessment:

To detect differences among three dMMR subtypes in terms of 3-year DFS and OS, a power analysis (Cohen's f = 0.25, α = 0.05, power = 80%) indicates a need for at least 122 dMMR patients. Assuming a dMMR prevalence of 8-15% and factoring in a 10% dropout rate, the total sample size is set at 1,500 patients.

-

Registry Quality and Data Management Plan (if registry or similar infrastructure is used):

* Data Validation & Quality Assurance:

A centralized data monitoring team will oversee data quality. Double entry and logic checks will be applied to ensure internal consistency, and site investigators will be asked to verify a random subset of submitted data.

* Source Data Verification:

Data will be cross-checked with local hospital records or pathology databases, particularly for key variables like MSI status, protein loss, and survival endpoints.

* Data Dictionary:

A comprehensive data dictionary will define each variable, data source, coding conventions (e.g., WHO-DD or MedDRA), and applicable clinical thresholds (e.g., tumor size cutoffs, lymph node positivity).

* Standard Operating Procedures (SOPs):

SOPs will be established for:

* Patient recruitment and consent
* Data entry and verification
* Histopathologic data review
* MSI/MMR testing techniques
* Management of missing or ambiguous data
* Adverse event reporting (if applicable)
* Periodic internal audits
* Plan for Missing Data:

Incomplete entries will be flagged and queried back to the site. Predefined rules will classify data as "missing," "not applicable," or "unavailable." Imputation will not be used for primary endpoints.

* Statistical Analysis Plan:

Descriptive statistics will summarize the distribution of dMMR and MSI status by tumor localization and other clinicopathological factors. Chi-square or Fisher's exact test will compare categorical variables.

* Kaplan-Meier curves and log-rank tests will compare DFS and OS between subtypes.
* Multivariable Cox regression models will adjust for confounders such as age, sex, stage, and treatment modality.
* MSI reporting frequency in biopsy specimens will be expressed as percentages and evaluated by hospital characteristics.

Dissemination Plan:

Study results will be submitted to national and international congresses and peer-reviewed journals. Aggregated, de-identified datasets may be shared upon request with institutional permission.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone curative-intent surgery for colon adenocarcinoma between June 1, 2025, and May 31, 2026 Surgery performed at a center with >30 colon cancer surgeries per year Availability of MMR protein immunohistochemistry (IHC) and/or MSI test results from resection specimen and/or preoperative endoscopic biopsy Signed informed consent for participation and data collection

Exclusion Criteria:

Non-adenocarcinoma malignancies of the colon (e.g., neuroendocrine tumors, lymphomas) Rectal cancers (defined as tumors within 15 cm of the anal verge on endoscopy or MRI) Incomplete medical or pathological records preventing classification of MMR status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from multiple high-volume general surgery centers across Turkey, including both public and private hospitals. The study will include institutions from major urban regions,as well as selected regional hospitals with established colorectal surgery programs.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and Anatomical Distribution of dMMR in Colon Cancer in Turkey | Within 30 days post-operative based on final pathology report
  The proportion of colon cancer patients with mismatch repair deficiency (dMMR), stratified by tumor location (right-sided vs left-sided colon). This will be determined using immunohistochemical analysis of MMR protein expression (MLH1, PMS2, MSH2, MSH6) in resection specimens.

SECONDARY OUTCOMES:
Frequency of MSI Reporting in Preoperative Endoscopic Biopsies | At time of initial diagnostic biopsy (baseline)
  The percentage of colon cancer cases in which MSI status is documented in the preoperative endoscopic biopsy pathology report. The goal is to evaluate the current national practice of early MSI testing prior to definitive surgery.
Three-Year Disease-Free Survival (DFS) and Overall Survival Across MMR Subtypes | 3 years from date of surgery
  Comparison of 3-year disease-free survival (DFS) among patients with MLH1/PMS2 loss, MSH2/MSH6 loss, and pMMR (sporadic) tumors. DFS is defined as the time from surgery to the first recurrence, metastasis, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Rencüzoğulları, Professor, Study Director — Koç University; Mustafa Öncel, Professor, Study Chair — İstanbul Medipol University; Burak Yavuz, M.D., Principal Investigator — Republic of Türkiye Ministry of Health Kozan State Hospital; Atıf Tekin, M.D., Principal Investigator — İstanbul Medipol University; Cihangir Akyol, Professor, Study Chair — Ankara University
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Medipol University, Istanbul
  - Koç University, Istanbul

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to confidentiality regulations and ethical considerations. Aggregated, de-identified data may be available upon reasonable request to the principal investigator, subject to institutional and ethical approval.

REFERENCES:
- [Background] de Gooyer PGM, Verschoor YL, van den Dungen LDW, Balduzzi S, Marsman HA, Geukes Foppen MH, Grootscholten C, Dokter S, den Hartog AG, Verbeek WHM, Woensdregt K, van den Broek JJ, Oosterling SJ, Schumacher TN, Kuhlmann KFD, Beets-Tan RGH, Haanen JBAG, van Leerdam ME, van den Berg JG, Chalabi M. Neoadjuvant nivolumab and relatlimab in locally advanced MMR-deficient colon cancer: a phase 2 trial. Nat Med. 2024 Nov;30(11):3284-3290. doi: 10.1038/s41591-024-03250-w. Epub 2024 Sep 15. PMID 39278994
- [Background] Anderson CE, Liska D. Treatment of Microsatellite-Unstable Rectal Cancer in Sporadic and Hereditary Settings. Clin Colon Rectal Surg. 2023 Aug 11;37(4):233-238. doi: 10.1055/s-0043-1770717. eCollection 2024 Jul. PMID 38882941